CLINICAL TRIAL: NCT02819895
Title: PRIMM Trial (Phone Reminder for IMMunization) in Ondo State, Nigeria
Brief Title: PRIMM Trial (Phone Reminder for IMMunization)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 15-012572
Record Dates: First submitted 2016-06-24; First posted 2016-06-30 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Immunization
Keywords: Phone Appointment Reminder; Immunization Rates; mHealth

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Parents of healthy newborn infants delivered at Mother and Child Hospital Ondo (Akure or Ondo), who live in Akure or Ondo Town and plan to receive their immunizations at MCH Ondo will receive their usual care (an immunization card). In addition they will received automated text, calls and emails (if applicable) reminders through a customized windows® software application when their child's immunization visit is due.
  Interventions: Other: A customized windows® software application
- Control (No Intervention): Parents of healthy newborn infants delivered at Mother and Child Hospital Ondo (Akure or Ondo), who live in Akure or Ondo Town and plan to receive their immunizations at MCH Ondo will receive usual care (an immunization card)

INTERVENTIONS:
Other: A customized windows® software application — A customized windows® software application with the ability to send automated voice call, SMS and email reminder about due dates for childhood routine immunizations.
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine if in a rural setting of Ondo State, Nigeria, a customized automated telephone and email immunization reminder system will be feasible, acceptable, and significantly improve immunization utilization rates.

DETAILED DESCRIPTION:
Background: Worldwide, vaccine preventable diseases account for 29% of all deaths between 1 month and 5 years, underscoring the importance of immunizations. In Nigeria, routine childhood immunization rates are unacceptably inconsistent and low, ranging from 35-85% at 14 weeks and 10-37% for all routine immunizations at 12-24 months.

GAP: The feasibility, acceptability and utility of an automated phone immunization reminder system have never been explored in this rural setting of Nigeria.

HYPOTHESIS: Given ~90% of the adult population in Nigeria uses a mobile phone, a customized mHealth immunization reminder system will be feasible and acceptable; and will significantly improve immunization rates in this rural setting of Ondo State, Nigeria.

METHODS: A prospective randomized controlled trial study design will be utilized. This study will recruit parents of healthy newborn infants delivered at Mother and Child Hospital Ondo, who live in Akure or Ondo Town and plan to receive their immunizations at Mother and Child Hospital Ondo.

DATA ANALYSIS: The proportion of immunization visits between intervention and control groups will be compared using a two-sided, two sample test of proportions with p <0.05 being significant. Secondary analysis will focus on the predictive value of social demographic variables on immunization rates.

ELIGIBILITY:
Inclusion Criteria:

1. Parents of healthy infants who have a cellular phone
2. Born at Mother and Child Hospital Ondo (Akure or Ondo Town)
3. Plans to receive immunizations at Mother and Child Hospital Ondo

Exclusion Criteria:

1. Parents of infants requiring hospital admission due to illness or prematurity.
2. Parents without a cellular phone

Ages: 1 Day to 1 Week | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Immunization Rates at 14 weeks | 14 Weeks
  To determine if an automated customized telephone and email immunization reminder system can increase the 14-week immunization rates, by at least 10% among those who receive immunization reminders versus those who do not.

SECONDARY OUTCOMES:
Immunization Rates at 14 Months | 14 Months
  To determine the effect of an automated customized phone and email immunization reminder system on the proportion of children completely immunized at 14 months among those who receive immunization reminders versus those who do not.
Timeliness of Immunization Receipt | 14 Months
  To determine if the proportion of infants who receive their immunizations within 1-week of its due date is higher in infants of parents who receive phone and email immunization reminders versus those who do not.

CONTACTS AND LOCATIONS:
Overall Officials: Osayame Ekhaguere, MBBS, MPH, Principal Investigator — Children's Hospital of Philadelphia; Andrew Steenhoff, MBBCh, Study Director — Children's Hospital of Philadelphia; Elizbeth Lowenthal, MD, MSCE, Study Director — Children's Hospital of Philadelphia
Locations (2):
- Nigeria (2):
  - Mother and Child Hospital Ondo, Akure, Ondo State
  - Mother and Child Hospital Ondo, Ondo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ekhaguere OA, Oluwafemi RO, Badejoko B, Oyeneyin LO, Butali A, Lowenthal ED, Steenhoff AP. Automated phone call and text reminders for childhood immunisations (PRIMM): a randomised controlled trial in Nigeria. BMJ Glob Health. 2019 Apr 3;4(2):e001232. doi: 10.1136/bmjgh-2018-001232. eCollection 2019. PMID 31139442